CLINICAL TRIAL: NCT03391778
Title: Long-Term Follow-Up (LTFU) of Participants Treated With ADP Adoptive Cell Therapies
Brief Title: Adoptive Cell Therapy Long-term Follow-up (LTFU) Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 208750; ADP-0000-002 (Other: Adaptimmune Therapeutics)
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-02

CONDITIONS: Neoplasms
Keywords: Long Term Follow Up; Adoptive Cell Therapy; Replication Competent Lentivirus
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants receiving ADP adoptive cell therapy (Experimental)
  Interventions: Biological: ADP adoptive cell therapy

INTERVENTIONS:
Biological: ADP adoptive cell therapy — No study drug is administered in this study. Participants who received ADP adoptive cell therapy in a previous trial will be evaluated in this trial for long-term safety and efficacy.

SUMMARY:
This trial will evaluate long term safety of participants who have received AdaptImmune (ADP) adoptive cell therapy for up to 15 years following last adoptive cell therapy infusion.

DETAILED DESCRIPTION:
Participants who received a ADP adoptive cell therapy will be enrolled in this non-therapeutic, multi-center, long term follow-up (LTFU) study and will be followed for up to 15 years post-infusion of lentiviral vector-based adoptive cell therapy. Participants will be monitored for safety following last adoptive cell therapy infusion.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have received at least one dose of ADP adoptive cell therapy agent.
* Participants who have completed ADP sponsored or supported interventional study or have withdrawn from it.
* Participants who have completed treatment as part of managed access to a GSK adoptive cell therapy.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* The investigator is responsible for review of medical history.
* Capable of giving signed informed consent.

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2032-04-01 (Estimated); Study Completion 2032-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with delayed adverse events (AEs) and serious adverse events (SAEs) | 15 years post last treatment
  AEs will be collected.

SECONDARY OUTCOMES:
Number of participants with Vesicular Stomatitis Virus G protein (VSV-G) Deoxyribonucleic acid (DNA) copies in peripheral blood samples | 15 years
  Peripheral blood samples will be collected for the assessment of VSV-G DNA copies.
Number of participants with Woodchuck hepatitis virus post-transcriptional regulatory element (WPRE) or Psi DNA copies in peripheral blood samples. | 15 years
  Peripheral blood samples will be collected for the assessment of WPRE or Psi DNA.
Number of participants with integrated vector sequences and vector integration patterns identified in peripheral blood samples | 15 years
  Peripheral blood samples will be collected for the assessment of Integrated vector sequences and vector integration patterns (e.g., polyclonal, oligoclonal, or monoclonal).
Number of deaths | 15 years
  Number of deaths will be summarized.
Time to death | 15 years
  Time to death will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Adaptimmune, Study Director — Adaptimmune
Locations (24):
- United States (13):
  - Emory University School of Medicine, Atlanta, Georgia
  - ADP Investigational Site, Baltimore, Maryland
  - National Cancer Institute - Center for Cancer Research, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center - New York, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) Hillman Cancer Center, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital, Milwaukee, Wisconsin
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
- Germany (2):
  - Klinikum rechts der Isar der Technischen Universität München, Munich, Bavaria
  - Uniklinik Köln, Cologne, North Rhine-Westphalia
- Fondazione IRCCS - Istituto Nazionale dei Tumori, Milan, Lombardy, Italy
- Antoni Van Leeuwenhoek Ziekenhuis, Amsterdam, Netherlands
- Hospital Universitario Virgen del Rocío, Seville, Spain
- United Kingdom (3):
  - University College London Hospitals NHS Foundation Trust, London
  - ADP Investigational Site, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: No